CLINICAL TRIAL: NCT04465721
Title: New York TREAT (Time Restricted EATing) to Improve Cardiometabolic Health Study
Brief Title: TREAT to Improve Cardiometabolic Health
Acronym: NY-TREAT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: New York University (Other); Salk Institute for Biological Studies (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Blandine Laferrere, Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AAAS7791; R01AG065569 (NIH)
Record Dates: First submitted 2020-07-01; First posted 2020-07-10 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Overweight and Obesity; Prediabetes
Keywords: Overweight; Obesity; Metabolic syndrome; Time restricted eating; Diabetes; Prediabetes; Lifestyle intervention; Smartphone app
MeSH Terms: conditions — Overweight; Obesity; Prediabetic State; Metabolic Syndrome; Intermittent Fasting; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Metabolically unhealthy mid-life adults with overweight or obesity who habitually eat for more than 13h/day, will be randomized to a restricted eating window to 10h/d (TRE group) or to their habitual eating window (≥ 13h, HABIT group), and followed up to 12 months.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HABIT Group (Active Comparator): Participants randomized to the HABIT group will maintain their habitual eating schedule (≥13-h).
  Interventions: Behavioral: HABIT
- TRE Group (Experimental): Participants randomized to TRE will reduce their eating window to a self-selected eating window (≤10-h).
  Interventions: Behavioral: TRE

INTERVENTIONS:
Behavioral: TRE — The TRE intervention will be administered and monitored via the study app. It combines self-monitoring behavior, daily eating window reminders, positive reinforcement based on number of log entries or based on meeting eating widow target, and basic lifestyle text messages. It also allows research staff to monitor in real-time, via the backend cloud, adherence to self-monitoring, and to reducing the eating window.
  Arms: TRE Group
Behavioral: HABIT — The HABIT intervention will be administered and monitored via the study app. It combines self-monitoring behavior, positive reinforcement based on number of log entries, and basic lifestyle text messages. It also allows research staff to monitor in real-time, via the backend cloud, adherence to self-monitoring.
  Arms: HABIT Group

SUMMARY:
Over half of American adults have overweight or obesity and are at high risk of developing type 2 diabetes and cardiovascular diseases. Although caloric restriction has many health benefits, it is difficult to sustain overtime for most people. Time restricted eating (TRE), a novel type of intermittent fasting, facilitates adherence to the intervention and results in weight loss and improvement of metabolism. The investigators propose to examine the efficacy of self-monitoring and TRE (10-h/d) vs. self-monitoring and habitual prolonged eating duration (HABIT) (13 hours/d) on weight loss and body composition, metabolic function and circadian biology, in metabolically unhealthy adults aged 50 to 75 y old, with overweight or obesity. The investigators hypothesize that TRE, compared to habitual long duration of eating, will decrease cardiovascular risk burden.

DETAILED DESCRIPTION:
American adults have a high prevalence of overweight, obesity and prediabetes. Small weight loss delays the progression to type 2 diabetes and decrease cardiovascular risk, yet adherence to long term calorie restriction is difficult to sustain. There is an urgency to find effective, easy-to implement and sustain, and affordable life style interventions. Restricting the food intake interval, or time restricted eating (TRE) has been shown in small-scale pilot studies to result in weight loss and improve metabolism, while being less challenging than calorie count. We propose to rigorously assess the efficacy and sustainability of self-monitoring with and without TRE, administered via a smartphone application, on weight loss and decreased cardiovascular risk. To achieve this goal, metabolically unhealthy mid-life adults with overweight or obesity who habitually eat for more than 13h/day, will be randomized to a self monitoring and restricted eating window to 10h/d (TRE) or to a self-monitoring and habitual eating window (13h, HABIT), and followed up to 12 months. Ambulatory measures of food intake, sleep, physical activity and glucose, and outpatient well controlled studies will be done to determine the effect of TRE versus habitual eating duration (HABIT), as well as the mediators of these effects. Hypotheses: 1) TRE vs. HABIT will result in decreased fat mass, measured by quantitative magnetic resonance, and effect mediated via decreased daily total energy intake, measured by double labeled water; 2) TRE vs. HABIT will result in lower insulin resistance, lower glycemia and shift in fuel utilization preferentially to lipid mobilization; 3) Adherence to the TRE intervention will be associated with greater weight loss at 3 months and weight maintenance at 12 months. Results from this study will provide important insights into understanding the physiological and molecular interactions between restricting daily eating interval and metabolic function, and could provide evidence for using TRE interventions to improve metabolic health and decrease cardiovascular risk in the large number of mid-life and older Americans in great need of life style intervention.

ELIGIBILITY:
Inclusion Criteria:

* age: 50-75y old
* BMI ≥25 and ≤45 kg/m2
* a diagnosis of prediabetes AND/OR fasting glucose 100 mg/dL and/or HbA1c 5.7% OR Type 2 Diabetes diet-controlled and/or treated with metformin AND meeting 2 or more of the following metabolic syndrome criteria:

  * diagnosis of hypertension on stable medication regimen
  * blood pressure >120/>80 mmHg
  * A diagnosis of dyslipidemia on stable regimen
  * triglycerides 150 mg/dL
  * HDL cholesterol men <40 mg/dL and women <50 mg/dL
  * waist circumference men: >102 cm (>40 in); women >88 cm (>35 in)
* in possession of a smart phone (iPhone or Android)
* 70% of days with logging adherence (2 or more log entries/day separated by at least 5h)
* Sleep duration 6-h, with habitual self-reported wake up time >5AM and before 11 AM and average self reported bed time <2AM
* habitually eat breakfast
* with weight stability within 5% of screening for the last 3 months
* English speaking (the App has not yet been translated)
* must live in the New York City metro area

Exclusion criteria:

* sleep disorder, e.g. known obstructive sleep apnea (OSA) on CPAP, severe OSA with apnea-hypopnea index >30 events/h, significant daytime symptoms of OSA, periodic limb movements of sleep, narcolepsy, current shift work or in last 6-mo, travel more than 1 time zone during intervention; severe insomnia with score 15 on Insomnia Severity Index
* significant organ system dysfunction/disease: severe pulmonary, kidney or cardiovascular disease; evidence of active illness (e.g., fever)
* history of seizure disorder
* previous bariatric surgery or on weight loss medication
* history of or current significant food intake or psychiatric disorder
* use of dietary supplements and/or medications known to affect sleep, circadian rhythms or metabolic function
* smoking tobacco or using illegal or recreational drugs
* consume excessive alcohol (women: >14 drinks/wk; men: >21 drinks/wk)
* anemia (hemoglobin <10 g/dl and hematocrit <30%)
* have conditions that render individual unable to complete all testing procedures [e.g., unable to stay overnight or frequent travel across 1 time zones]
* extreme early and late chronotypes (> 2AM bed time and wake up time before 5AM and > 11AM)
* severe food allergies
* unwilling/unable to provide informed consent

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Fat mass | 0, 3, and 12 months
  Changes in fat mass (kg) will be measured by quantitative magnetic resonance (QMR) on day 0 and day 13 of ambulatory assessments at the 0 and 3 month study period, and again at 12 months.
Energy intake | 0, 3 months
  Energy intake (EI) will be calculated from total daily energy expenditure (EE) measured by doubly labeled water (DLW), and changes in body energy stores (ΔES), measured by QMR over the 2-wk ambulatory assessments of the 0 and 3 month study periods: EI (kcal/d) = EEDLW + ΔES.
Body weight | 0, 3, 12 months
  Changes in body weight (kg) will be measured to the nearest 0.01 kg with a digital scale at 0 and 3 months, and again at 12 months.
Insulin resistance (HOMA-IR) | 0, 3, 12 months
  Fasting serum insulin and plasma glucose concentrations will be used to calculate changes in insulin resistance (HOMA-IR): [fasting insulin (mU/mL) x fasting glucose (mmol/L)]/22.5 at 0 and 3 months, and again at 12 months.
Glucose levels | 0, 3,12 months
  Glucose changes will be assessed by the total and incremental 24-hour glucose AUC, from ambulatory CGM at 0 and 3 months.
Glucose variability | 0, 3,12 months
  CGM data will be used to calculate standard measures of glucose variability (GV), including mean amplitude of glycemic excursion (MAGE) changes at 0 and 3 months.
Sleep assessment | 0, 3,12 months
  Sleep duration will be assessed by changes in bedtime, waketime, and total sleep time, recorded by actigraphy during the 2-wk ambulatory assessments at 0, 3, and 12 months.
Adherence | 0, 3,12 months
  Adherence will be assessed by % of days with at least 2 or more entries logged at least 5h apart/day

SECONDARY OUTCOMES:
Diet composition by ASA24 | 0, 3, 12 months
  % of carbs, fat and protein in diet by ASA24 on 3 non-consecutive days (2 weekdays and one weekend day) during each ambulatory assessment and during the 3 months intervention.
Matsuda Index (Insulin resistance) | 0, 3 months
  Fasting and OGTT glucose and insulin levels are used to calculate the Matsuda index:
  10,000/([fasting insulin (mU/mL)x fasting glucose (mmol/L)]x [mean OGTT insulin (mU/mL) x mean OGTT glucose (mmol/L)])
Insulinogenic Index | 0, 3 months
  Calculated by the AUC insulin/AUC glucose during OGTT.
Free fatty acids (FFA) | 0, 3, 12 months
  Measured from a fasting blood sample
Ketones | 0, 3, 12 months
  The concentration of ketones (beta-OH-butyrate) will be measured from a fasting blood sample.
Physical activity | 0, 3, 12 months
  Assessed by step count during 14 day ambulatory assessment periods at 0,3, and 12 months.
Inflammation markers | 0, 3, 12 months
  Measured from a fasting blood sample.
Oxidative stress | 0, 3, 12 months
  Measured from a fasting blood sample
Lipid profile | 0, 3, 12 months
  Measured from a fasting blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Blandine Laferrère, M.D., Ph.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Columbia University is committed to the open and timely dissemination of research outcomes. Investigators in this proposed project are aware of and agree to abide by the principles for sharing research resources, as described by NIH in "Principles and Guidelines for Recipients of NIH Research Grants and Contracts on Obtaining and Disseminating Biomedical Research Programs." All data used in this proposal will de-identified, and accessed using a secure data area using a shared drive, protected by password only to be accessed by those directly involved in the clinical research. All transfer of data will use encrypted methods. Wherever applicable, fully de-identified data will be deposited to appropriate public repositories, following the Federal Health Insurance Privacy and Portability Act (HIPAA).
Time Frame: This will occur no longer than 6 months after publications of the data generated by this application, or, 18 months after completion of the funding period, should no data had been published.
Access Criteria: The data generated in this grant will be presented at national or international conferences and published in a timely fashion. All final peer-reviewed manuscripts that arise from this proposal will be submitted upon acceptance for publication to the digital archive NIH National Library of Medicine PubMed Central (PMC) database, according to the NIH Policy on Enhancing Public Access to Archived Publications Resulting from NIH Funded Research. Any data released for publication will be for research purposes only and will not include identifiable data on any of the participants.

REFERENCES:
- [Derived] Santos-Baez LS, Ravelli MN, Diaz-Rizzolo DA, Popp CJ, Gallagher D, Cheng B, Schoeller D, Laferrere B. Dietary misreporting: a comparative study of recalls vs energy expenditure and energy intake by doubly-labeled water in older adults with overweight or obesity. BMC Med Res Methodol. 2025 Apr 26;25(1):115. doi: 10.1186/s12874-025-02568-4. PMID 40287632
- [Derived] Diaz-Rizzolo DA, Santos Baez LS, Popp CJ, Borhan R, Sordi-Guth A, Manoogian ENC, Panda S, Cheng B, Laferrere B. Late eating is associated with poor glucose tolerance, independent of body weight, fat mass, energy intake and diet composition in prediabetes or early onset type 2 diabetes. Nutr Diabetes. 2024 Oct 25;14(1):90. doi: 10.1038/s41387-024-00347-6. PMID 39455572
- [Derived] Metzendorf MI, Wieland LS, Richter B. Mobile health (m-health) smartphone interventions for adolescents and adults with overweight or obesity. Cochrane Database Syst Rev. 2024 Feb 20;2(2):CD013591. doi: 10.1002/14651858.CD013591.pub2. PMID 38375882
- [Derived] Santos-Baez LS, Garbarini A, Shaw D, Cheng B, Popp CJ, Manoogian ENC, Panda S, Laferrere B. Time-restricted eating to improve cardiometabolic health: The New York Time-Restricted EATing randomized clinical trial - Protocol overview. Contemp Clin Trials. 2022 Sep;120:106872. doi: 10.1016/j.cct.2022.106872. Epub 2022 Aug 4. PMID 35934281